CLINICAL TRIAL: NCT05666791
Title: The Association Between Diabetes Stress, Self-efficacy, Self-management, and Glycemic Control in Children and Adolescents With Type 1 Diabetes Mellitus
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202210117RINC
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Children and Adolescents With Type 1 Diabetes Mellitus
Keywords: Children and adolescents with type 1 diabetes mellitus, Diabetes stress, Self-efficacy, Self-management, HbA1c

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aims of this study were to: (1) Investigate the association between perceived diabetes-specific stress, self-efficacy, self-management and glycemic control in children and adolescents with type 1 diabetes mellitus (T1D). (2) Explore whether self-efficacy and self-management mediates the relationship between perceived diabetes stress and glycemic control in adolescents with type 1 diabetes (T1D). (3) Explore whether self-efficacy and self-management moderated the relationship between perceived diabetes stress and glycemic control in adolescents with type 1 diabetes (T1D).

DETAILED DESCRIPTION:
Investigators have found that type 1 diabetes mellitus (T1D) is more commonly diagnosed in childhood compared with adulthood; optimizing HbA1c level is essential for reducing the risk and severity of complications; childhood glycemic control is also associated with further risk of physical and psychological health problems as an adult, nevertheless, adolescence is a stage of transition to adulthood, compared with other age groups, and adolescents with type 1 diabetes mellitus (T1D) have worse glycemic control.

Diabetes-specific stress has been previously defined as a negative experience involving physiological, emotional, and behavior changes in relation to a diabetes specific stressor, it is also associated with psychological well-being and mediates the relationship between diabetes-specific cognitive appraisals and glycemic control.

Cross-sectional studies also indicate that self-efficacy and self-management are positively correlated, importantly, in adolescents with type 1 diabetes mellitus (T1D), higher self-efficacy was associated with lower HbA1c levels; higher self-efficacy was also directly associated with better self-management and lower HbA1c levels.

Individuals with type 1 diabetes mellitus (T1D) need to self-manage their HbA1c levels throughout their lives, self-management also refers to the daily active management of illness-related activities for achieving glycemic control; accordingly, self-management in adolescents is always challenging, and glycemic control is typically at its worst in the transitional period between adolescence and adulthood.

Considering that diabetes-specific stress might be directly associated with self-efficacy, self-management and glycemic control in children and adolescents with type 1 diabetes mellitus (T1D), further study is still warranted. Understanding the factors and pathways associated with subsequent HbA1c levels could assist in the development of comprehensive and timely interventions to improve glycemic control among this population.

This study applied as a cross-sectional study; Demographic characteristics, Diabetes-specific stress, self -efficacy and self-management were collected using self -reported questionnaires; HbA1c levels will be obtained from medical records.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were having had a diagnosis of type 1 diabetes mellitus for more than 6 months, screened and referred by a pediatric endocrinology physician, being aged 8~25 years old, and also being able to read or communicate verbally in mandarin Chinese.

Exclusion Criteria:

* Participants diagnosed with cognitive or mental health problems were excluded.

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with type 1 diabetes mellitus being treated at NTUH will be recruited. The inclusion criteria were having had a diagnosis of type 1 diabetes mellitus for more than 6 months, screened and referred by a pediatric endocrinology physician, being aged 8~25 years old, and also being able to read or communicate verbally in mandarin Chinese.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-21 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Demographic characteristics | 5 minutes
  Demographic characteristics include participants' age, gender, diabetes treatment plan, body high and body weight; caregiver's age, income, education background, occupation and health condition.
Diabetes specific-stress | 10 minutes
  The 24-item Diabetes Stress Questionnaire-short form (DSQ-SF) demonstrated good internal consistency and convergent validity; it's also a quick, cost-effective and useful tool for measuring perceived stress in youth with type 1 diabetes mellitus; higher scores indicating higher levels of diabetes specific-stress.
Self-management | 10 minutes
  The 23-item Short Form Chinese version of the Self-Management of Type 1 Diabetes for Adolescents Scale (C-SMOD-A-23) was used to assess patient collaboration with parents; patient diabetes care activities, problem-solving behaviors and communication, and healthy lifestyle goals; the higher the item mean score, the greater the patient's self-management ability.
Self-efficacy | 5 minutes
  The 10-item Chinese version of the self-efficacy scale was used to measure self-confidence in facing potential challenges in diabetes self-management in children and adolescents with Type 1 Diabetes; the higher the item mean score, the higher the patient's self-efficacy.

IPD SHARING:
Plan to Share IPD: Undecided